CLINICAL TRIAL: NCT00733304
Title: An Extension Study to Protocol MD7108240: Pazopanib Eye Drops in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: An Extension to Study MD7108240
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD7111396
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Macular Degeneration
Keywords: age-related macular degeneration (AMD); choroidal neovascularization (CNV); vascular endothelial growth factor (VEGF); pazopanib; angiogenesis
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 5 mg/ml TID (Experimental): eligible participants received 5 mg/ml Pazopanib eye drops three times daily (TID)
  Interventions: Drug: Pazopanib
- 2 mg/ml TID (Experimental): eligible participants received 2 mg/ml Pazopanib eye drops three times daily
  Interventions: Drug: Pazopanib
- 5 mg/ml QD (Experimental): eligible participants received 5 mg/ml Pazopanib eye drops once daily (QD)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 5 mg/ml TID, 2 mg/ml TID or 5 mg/ml QD

SUMMARY:
This is a two month study to allow continued treatment with pazopanib eye drops. Study may be extended to 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in Phase IIa study MD7108240 and who did not experience AMD disease progression requiring rescue therapy during pazopanib treatment or require discontinuation of pazopanib eye drops for safety reasons
* Best-corrected ETDRS visual acuity in the study eye of 23 letters (20/320 or 4/63) or better at screening.
* QTcB or QTcF < 450msec; or QTc < 480msec in subjects with Bundle Branch Block.
* Subject is willing and able to return for all study visits, and is willing and able to comply with all protocol requirements and procedures.
* Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. If the subject is unable to read the consent form due to visual impairment then the consent must be read to the subject verbatim by person administering the consent, a family member or legally acceptable representative. If the subject is unable to provide written informed consent due to visual impairment, then written informed consent on behalf of the subject must be provided by a legally acceptable representative. (Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations and ethics committee policy.)

Exclusion Criteria:

* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation of the fundus for photographs, fluorescein angiography and OCT.
* Vitreous, subretinal or retinal hemorrhage in the study eye that is unrelated to AMD.
* Intraocular surgery in the study eye within 3 months of dosing.
* Use of topical ocular medications (other than pazopanib) in the study eye within 7 days of first dose of investigational product or expected use of topical ocular medications during the treatment period, with the exception of artificial tears.
* Current use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol).
* An unwillingness to refrain from wearing contact lenses starting from the screening visit, through the follow-up visit
* ALT or AST above the upper limit of normal or total bilirubin ≥ 1.5 times the upper limit of normal at baseline. Note: Laboratory tests outside of the normal range may be repeated at the discretion of the Investigator.
* Medical history or condition:
* Uncontrolled Diabetes Mellitus, with hemoglobin A1c (HbA1c) > 10%.
* Myocardial infarction or stroke within 6 months of screening.
* Active bleeding disorder.
* Major surgery within 1 month of screening.
* Hepatic impairment.
* Uncontrolled hypertension, based on criteria provided in the protocol. Note: Initiation or adjustment of antihypertensive medications is permitted prior to study entry provided the referenced criteria are met.
* Use of prohibited medications listed in the protocol within the restricted timeframe relative to the first dose of study medication.
* A condition or situation which, in the opinion of the investigator, may result in significant risk to the subject, confound the study results or interfere significantly with participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06-25 (Actual); Primary Completion 2009-09-09 (Actual); Study Completion 2009-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (8):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Salt Lake City, Utah
- Australia (3):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Italy (4):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an extension study to protocol MD7108240 (NCT00612456). It was a multi-center, double-masked, randomized, parallel-group dose-ranging study of repeat topical ocular doses of pazopanib from 25 June 2008 to 9 September 2009. The study was conducted in 14 centers in the United States, Italy, and Australia.
Pre-assignment Details: Randomized participants without progression of age-related macular degeneration (AMD) and/or requiring rescue therapy during the 28-day treatment period in study MD7108240 (NCT00612456) were included in this study. A total of 42 participants were randomized in the study.
Groups:
- 5 mg/mL TID: Eligible participants received 5 milligram/milliliter (mg/mL) Pazopanib eye drops three times daily for a treatment period of five months.
- 2 mg/mL TID: Eligible participants received 2 mg/mL Pazopanib eye drops three times daily for a treatment period of five months.
- 5 mg/mL QD: Eligible participants received 5 mg/mL Pazopanib eye drops once daily for a treatment period of five months.
Period: Overall Study
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Started | 19 | 15 | 8
Completed | 12 | 12 | 3
Not Completed | 7 | 3 | 5
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 3 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5 mg/mL TID: Eligible participants received 5 mg/mL Pazopanib eye drops three times daily for a treatment period of five months.
- Total: Total of all reporting groups
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD | Total
Number analyzed (Participants) | 19 | 15 | 8 | 42
Age, Customized [Count of Participants; unit: Participants]
  55 to 88 aged | 19 | 15 | 8 | 42
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    Female | 15 | 7 | 5 | 27
    Male | 4 | 8 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 19 | 15 | 8 | 42
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Day 1) in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. SBP and DBP were recorded from Baseline up to 6 months. At screening and Baseline, if the single measured value of blood pressure was above 150 millimeters of mercury (mm Hg) systolic or 95 mm Hg diastolic, then blood pressure measurement could not be repeated. If, the SBP was <80 or >140 mm Hg and DBP was <40 or >90 mm Hg, then measurement of BP was repeated. Three consecutive blood pressure readings that were less than 150 mmHg systolic and 95 mmHg diastolic were taken with each measurement separated by at least 1 hour.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population included all participants who received at least one dose of the study drug. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Groups:
- 5 mg/mL TID: Eligible participants received 5 mg/mL Pazopanib eye drops three times daily for a treatment period of five months and were followed-up for 7-14 days after the last dose of the study drug.
- 2 mg/mL TID: Eligible participants received 2 mg/mL Pazopanib eye drops three times daily for a treatment period of five months and were followed-up for 7-14 days after the last dose of the study drug.
- 5 mg/mL QD: Eligible participants received 5 mg/mL Pazopanib eye drops once daily for a treatment period of five months and were followed-up for 7-14 days after the last dose of the study drug.
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Millimeters of mercury (mmHg)
  DBP, Month 1: number analyzed (Participants) | 19 | 14 | 8
  DBP, Month 1 | 3.5 (9.05) | -0.4 (8.40) | 1.1 (3.98)
  DBP, Month 2: number analyzed (Participants) | 18 | 13 | 8
  DBP, Month 2 | 1.8 (8.79) | 1.6 (8.32) | -0.5 (7.09)
  DBP, Month 3: number analyzed (Participants) | 15 | 12 | 4
  DBP, Month 3 | 3.9 (8.03) | -0.9 (8.16) | 1.5 (7.42)
  DBP, Month 4: number analyzed (Participants) | 12 | 11 | 5
  DBP, Month 4 | 0.0 (8.49) | -0.4 (6.09) | 0.0 (6.12)
  DBP, Month 5: number analyzed (Participants) | 12 | 12 | 3
  DBP, Month 5 | 8.6 (11.83) | 1.8 (7.40) | 4.7 (19.73)
  DBP, Follow-up: number analyzed (Participants) | 17 | 13 | 6
  DBP, Follow-up | 3.3 (9.04) | 1.8 (9.59) | -2.8 (11.11)
  SBP, Month 1: number analyzed (Participants) | 19 | 14 | 8
  SBP, Month 1 | -2.4 (10.55) | 0.5 (12.68) | -2.3 (9.22)
  SBP, Month 2: number analyzed (Participants) | 18 | 13 | 8
  SBP, Month 2 | -0.4 (14.91) | -3.0 (15.37) | -4.0 (7.91)
  SBP, Month 3: number analyzed (Participants) | 15 | 12 | 4
  SBP, Month 3 | -0.5 (16.29) | 1.8 (12.46) | 0.8 (10.63)
  SBP, Month 4: number analyzed (Participants) | 12 | 11 | 5
  SBP, Month 4 | -4.1 (10.37) | -1.9 (6.98) | -1.0 (8.83)
  SBP, Month 5: number analyzed (Participants) | 12 | 12 | 3
  SBP, Month 5 | 0.0 (17.16) | -1.3 (14.71) | -9.7 (1.15)
  SBP, Follow-up: number analyzed (Participants) | 17 | 13 | 6
  SBP, Follow-up | 0.6 (12.65) | 0.9 (13.44) | -2.3 (5.99)

2. Primary Outcome: Change From Baseline (Day 1) in Heart Rate Over Period
Description: Heart rate was measured over 6 months. Baseline value was recorded on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value. Heart rate measurement were repeated in case it was in range < 50 beats per minute (bpm) or >110 bpm.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
bpm
  Month 1: number analyzed (Participants) | 19 | 14 | 8
  Month 1 | -0.6 (9.81) | 2.4 (9.19) | 5.1 (9.82)
  Month 2: number analyzed (Participants) | 18 | 13 | 8
  Month 2 | -0.3 (8.50) | 1.3 (8.89) | 5.0 (9.52)
  Month 3: number analyzed (Participants) | 15 | 12 | 4
  Month 3 | 1.4 (10.92) | -2.5 (13.90) | 1.3 (7.37)
  Month 4: number analyzed (Participants) | 12 | 11 | 5
  Month 4 | -2.0 (9.80) | 0.7 (9.85) | -2.2 (8.90)
  Month 5: number analyzed (Participants) | 12 | 12 | 3
  Month 5 | -0.8 (7.70) | 0.6 (10.90) | 9.3 (20.03)
  Follow-up: number analyzed (Participants) | 17 | 13 | 6
  Follow-up | -0.2 (6.78) | -1.8 (8.07) | 5.0 (11.22)

3. Primary Outcome: Change From Baseline (Day 1) in Albumin and Hemoglobin Over Period
Description: Albumin and hemoglobin values were recorded at Baseline, Month2, and till follow-up (Month 6). Baseline was recorded on Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1), Month 2, 5 and approximately up to Month 6
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Grams per liter
  Albumin, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Albumin, Month 2 | 0.6 (1.46) | -0.7 (1.38) | -1.1 (1.96)
  Albumin, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Albumin, Month 5 | 0.3 (2.15) | -1.0 (1.34) | -3.0 (1.00)
  Albumin, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Albumin, Follow-up | -0.4 (1.67) | -1.1 (1.45) | 0.2 (1.30)
  Hemoglobin, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Hemoglobin, Month 2 | 2.1 (6.95) | -0.5 (4.22) | -1.3 (8.35)
  Hemoglobin, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Hemoglobin, Month 5 | -0.2 (10.04) | 0.3 (5.05) | -6.0 (0.00)
  Hemoglobin, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Hemoglobin, Follow-up | -0.2 (8.65) | 0.4 (8.66) | 2.5 (5.26)

4. Primary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferases (ALT), and Aspartate Aminotransferases (AST) Over Period
Description: ALP, ALT and AST values were measured over 5 months and till the follow-up period. Baseline value was recorded pre-dose Day 1. Change from Baseline is the value at indicated time point minus the Baseline value.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
International units per Liter (IU/L)
  ALP, Month 1: number analyzed (Participants) | 18 | 14 | 8
  ALP, Month 1 | -2.8 (8.01) | -0.6 (11.24) | -0.1 (5.94)
  ALP, Month 2: number analyzed (Participants) | 18 | 13 | 8
  ALP, Month 2 | 1.1 (7.73) | 1.8 (6.03) | -2.3 (8.31)
  ALP, Month 3: number analyzed (Participants) | 15 | 12 | 4
  ALP, Month 3 | 1.2 (8.19) | 1.3 (8.94) | -7.5 (5.92)
  ALP, Month 4: number analyzed (Participants) | 12 | 10 | 5
  ALP, Month 4 | 2.6 (10.58) | -3.5 (8.64) | -1.8 (6.91)
  ALP, Month 5: number analyzed (Participants) | 11 | 11 | 3
  ALP, Month 5 | 0.7 (10.82) | -1.6 (8.99) | 8.3 (13.80)
  ALP, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  ALP, Follow-up | 3.7 (13.77) | 0.1 (7.98) | 3.6 (4.62)
  ALT, Month 1: number analyzed (Participants) | 18 | 14 | 8
  ALT, Month 1 | 2.1 (3.80) | -0.1 (1.90) | -0.4 (3.93)
  ALT, Month 2: number analyzed (Participants) | 18 | 13 | 8
  ALT, Month 2 | 3.0 (3.41) | 2.0 (4.12) | 2.1 (4.94)
  ALT, Month 3: number analyzed (Participants) | 15 | 12 | 4
  ALT, Month 3 | 0.9 (5.54) | -0.7 (3.39) | -0.8 (3.59)
  ALT, Month 4: number analyzed (Participants) | 12 | 10 | 5
  ALT, Month 4 | 2.1 (5.07) | -1.3 (4.55) | -0.4 (2.30)
  ALT, Month 5: number analyzed (Participants) | 11 | 11 | 3
  ALT, Month 5 | 2.3 (3.23) | -2.2 (6.82) | -1.0 (3.00)
  ALT, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  ALT, Follow-up | 2.2 (4.07) | -1.1 (3.21) | -0.2 (2.17)
  AST, Month 1: number analyzed (Participants) | 18 | 14 | 8
  AST, Month 1 | 1.7 (3.16) | 0.0 (3.94) | -0.5 (3.78)
  AST, Month 2: number analyzed (Participants) | 18 | 13 | 8
  AST, Month 2 | 2.4 (3.42) | 1.6 (3.93) | 1.0 (2.93)
  AST, Month 3: number analyzed (Participants) | 15 | 12 | 8
  AST, Month 3 | 1.1 (3.94) | -1.0 (5.56) | 0.0 (2.16)
  AST, Month 4: number analyzed (Participants) | 12 | 10 | 8
  AST, Month 4 | 0.1 (3.18) | 0.0 (3.74) | 1.2 (2.39)
  AST, Month 5: number analyzed (Participants) | 11 | 11 | 8
  AST, Month 5 | 1.8 (3.16) | -1.4 (5.33) | 0.3 (2.89)
  AST, Follow-up: number analyzed (Participants) | 16 | 11 | 8
  AST, Follow-up | 2.0 (3.18) | -1.1 (3.78) | 1.2 (4.15)

5. Primary Outcome: Change From Baseline (Day 1) in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelets, and White Blood Cell Count Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. The above mentioned hematological parameters were recorded from Baseline up to 5 months.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Giga per Liter (G/L)
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Giga per Liter (G/L)
  Basophils, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Basophils, Month 2 | 0.008 (0.0246) | 0.008 (0.0157) | -0.003 (0.0271)
  Basophils, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Basophils, Month 5 | 0.007 (0.0237) | 0.006 (0.0168) | -0.010 (0.0141)
  Bsophils, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Bsophils, Follow-up | 0.010 (0.0234) | -0.003 (0.0142) | 0.00 (0.00)
  Eosinophils, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Eosinophils, Month 2 | -0.043 (0.1604) | 0.010 (0.1204) | -0.088 (0.1784)
  Eosinophils, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Eosinophils, Month 5 | 0.034 (0.0952) | -0.009 (0.1324) | 0.030 (0.1131)
  Eosinophils,Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Eosinophils,Follow-up | 0.046 (0.1623) | 0.007 (0.1083) | 0.032 (0.0613)
  Lymphocytes, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Lymphocytes, Month 2 | 0.077 (0.8534) | 0.051 (0.4203) | -0.031 (0.3855)
  Lymphocytes, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Lymphocytes, Month 5 | -0.004 (0.5848) | 0.068 (0.2245) | 0.130 (0.3536)
  Lymphocytes, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Lymphocytes, Follow-up | -0.058 (0.4984) | 0.090 (0.3412) | 0.062 (0.1959)
  Monocytes, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Monocytes, Month 2 | 0.025 (0.1304) | 0.025 (0.1621) | 0.020 (0.1812)
  Monocytes, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Monocytes, Month 5 | 0.006 (0.2047) | 0.036 (0.1272) | -0.015 (0.1202)
  Monocytes, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Monocytes, Follow-up | -0.035 (0.1506) | 0.002 (0.1293) | 0.030 (0.0942)
  Platelets, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Platelets, Month 2 | -1.1 (21.84) | 1.3 (21.39) | 11.9 (29.30)
  Platelets, Month 5: number analyzed (Participants) | 11 | 12 | 2
  Platelets, Month 5 | 1.3 (33.83) | -10.9 (15.48) | 70.0 (62.23)
  Platelets, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Platelets, Follow-up | -3.3 (22.50) | -7.3 (19.31) | 8.3 (7.50)
  White blood cells, Month 2: number analyzed (Participants) | 18 | 13 | 8
  White blood cells, Month 2 | -0.42 (1.986) | -0.02 (1.027) | 0.26 (1.334)
  White blood cells, Month 5: number analyzed (Participants) | 11 | 12 | 2
  White blood cells, Month 5 | -1.41 (2.938) | -0.00 (1.484) | 0.50 (1.697)
  White blood cells, Follow-up: number analyzed (Participants) | 16 | 12 | 4
  White blood cells, Follow-up | -0.89 (2.614) | 0.76 (2.558) | -0.07 (2.251)

6. Primary Outcome: Change From Baseline (Day 1) in Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Over here, the change is % Basophils at month x - % Basophils at Baseline. Baseline measurement was recorded at Day 1. Percentage change in the hematological parameter mentioned above was recorded from Baseline up to 5 months.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Percentage of cells
  % Basophils, Month 2: number analyzed (Participants) | 18 | 13 | 8
  % Basophils, Month 2 | 0.12 (0.340) | 0.12 (0.251) | -0.05 (0.293)
  % Basophils, Month 5: number analyzed (Participants) | 11 | 12 | 3
  % Basophils, Month 5 | 0.11 (0.274) | 0.08 (0.226) | -0.20 (0.173)
  % Basophils, Follow-up: number analyzed (Participants) | 16 | 12 | 5
  % Basophils, Follow-up | 0.17 (0.320) | -0.01 (0.193) | -0.04 (0.182)
  % Eosinophils, Month 2: number analyzed (Participants) | 18 | 13 | 8
  % Eosinophils, Month 2 | -0.44 (2.352) | 0.19 (1.366) | -1.08 (2.089)
  % Eosinophils, Month 5: number analyzed (Participants) | 11 | 12 | 3
  % Eosinophils, Month 5 | 0.60 (1.564) | 0.16 (1.879) | -0.30 (0.964)
  % Eosinophils,Follow-up: number analyzed (Participants) | 16 | 12 | 5
  % Eosinophils,Follow-up | 0.64 (2.601) | 0.04 (1.828) | -0.56 (4.245)
  % lymphocytes, Month 2: number analyzed (Participants) | 18 | 13 | 8
  % lymphocytes, Month 2 | 2.29 (11.781) | -0.52 (7.788) | -0.96 (4.260)
  % lymphocytes, Month 5: number analyzed (Participants) | 11 | 12 | 3
  % lymphocytes, Month 5 | 4.42 (9.734) | 0.83 (4.759) | 3.87 (8.051)
  % lymphocytes, Follow-up: number analyzed (Participants) | 16 | 12 | 5
  % lymphocytes, Follow-up | 2.29 (7.790) | -0.62 (4.021) | -3.66 (17.637)
  % monocytes, Month 2: number analyzed (Participants) | 18 | 13 | 8
  % monocytes, Month 2 | 0.57 (1.671) | 0.50 (1.974) | -0.19 (1.277)
  % monocytes, Month 5: number analyzed (Participants) | 11 | 12 | 3
  % monocytes, Month 5 | 1.24 (3.029) | 0.59 (1.358) | -0.67 (0.611)
  % monocytes, Follow-up: number analyzed (Participants) | 16 | 12 | 5
  % monocytes, Follow-up | 0.06 (1.803) | -0.32 (1.236) | 0.96 (3.247)
  %Total neutrophils, Month 2: number analyzed (Participants) | 18 | 13 | 8
  %Total neutrophils, Month 2 | -2.54 (12.125) | -0.28 (7.709) | 2.27 (3.593)
  %Total neutrophils, Month 5: number analyzed (Participants) | 11 | 12 | 3
  %Total neutrophils, Month 5 | -6.36 (12.291) | -1.65 (6.020) | -2.70 (7.826)
  %Total neutrophils, Follow-up: number analyzed (Participants) | 16 | 12 | 5
  %Total neutrophils, Follow-up | -3.16 (9.812) | 0.90 (5.801) | 3.30 (24.091)

7. Primary Outcome: Change From Baseline (Day 1) in Direct Bilirubin, Total Bilirubin, and Creatinine Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. Direct bilirubin, total bilirubin, and creatinine were recorded from Baseline up to 6 months
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Micromoles per Liter (umol/L)
  Direct bilirubin, Month 1: number analyzed (Participants) | 18 | 14 | 8
  Direct bilirubin, Month 1 | -0.1 (0.47) | -0.2 (0.58) | 0.3 (0.71)
  Direct bilirubin, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Direct bilirubin, Month 2 | 0.2 (0.92) | 0.0 (0.91) | 0.5 (0.93)
  Direct bilirubin, Month 3: number analyzed (Participants) | 15 | 12 | 4
  Direct bilirubin, Month 3 | -0.1 (0.64) | -0.5 (0.90) | 0.0 (0.0)
  Direct bilirubin, Month 4: number analyzed (Participants) | 12 | 10 | 5
  Direct bilirubin, Month 4 | -0.1 (0.51) | -0.1 (0.99) | 0.8 (1.10)
  Direct bilirubin, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Direct bilirubin, Month 5 | 0.1 (0.70) | -0.1 (0.70) | 0.0 (0.0)
  Direct bilirubin, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Direct bilirubin, Follow-up | -0.1 (1.00) | -0.2 (1.17) | 0.4 (0.89)
  Total bilirubin, Month 1: number analyzed (Participants) | 18 | 14 | 8
  Total bilirubin, Month 1 | -0.7 (3.98) | -1.4 (2.02) | 0.4 (2.26)
  Total bilirubin, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Total bilirubin, Month 2 | 0.3 (1.78) | 0.2 (2.70) | 0.5 (3.82)
  Total bilirubin, Month 3: number analyzed (Participants) | 15 | 12 | 4
  Total bilirubin, Month 3 | -1.2 (4.04) | -0.6 (2.50) | -2.0 (1.63)
  Total bilirubin, Month 4: number analyzed (Participants) | 12 | 10 | 5
  Total bilirubin, Month 4 | -0.3 (2.02) | -0.9 (1.52) | -0.4 (2.97)
  Total bilirubin, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Total bilirubin, Month 5 | -0.7 (2.28) | -0.5 (2.50) | -2.0 (2.00)
  Total bilirubin, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Total bilirubin, Follow-up | -1.1 (2.43) | 0.3 (2.97) | -0.8 (3.35)
  Creatinine, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Creatinine, Month 2 | 3.5 (9.65) | 3.0 (9.23) | -5.0 (7.07)
  Creatinine, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Creatinine, Month 5 | -0.5 (5.16) | 2.3 (5.44) | -6.0 (5.20)
  Creatinine, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Creatinine, Follow-up | 4.3 (8.65) | 3.5 (8.66) | -7.0 (14.46)

8. Primary Outcome: Change From Baseline in Calcium, Chloride, Carbon di Oxide Equivalent Content, Glucose, Potassium, Sodium, and Urea Blood Urea Nitrogen (BUN) Over Period
Description: Change from Baseline (Day 1) is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. Calcium, chloride, carbon di oxide equivalent content (CO2), glucose, potassium, sodium, and urea/blood urea nitrogen (BUN) was recorded from Baseline up to Follow-up.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Millimoles per Liter (mmol/L)
  Calcium, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Calcium, Month 2 | 0.000 (0.1006) | -0.020 (0.0840) | -0.050 (0.1189)
  Calcium, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Calcium, Month 5 | -0.006 (0.1105) | -0.045 (0.0934) | -0.100 (0.0917)
  Calcium, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Calcium, Follow-up | -0.026 (0.0902) | -0.010 (0.0542) | -0.028 (0.1221)
  Chloride, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Chloride, Month 2 | 0.1 (2.59) | -0.2 (1.99) | 0.5 (1.77)
  Chloride, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Chloride, Month 5 | -0.3 (2.45) | 0.5 (1.37) | -2.0 (1.73)
  Chloride, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Chloride, Follow-up | 0.0 (2.42) | 0.1 (1.70) | -0.2 (2.59)
  CO2, Month 2: number analyzed (Participants) | 18 | 13 | 8
  CO2, Month 2 | -0.4 (2.17) | -1.3 (2.14) | -1.3 (2.60)
  CO2, Month 5: number analyzed (Participants) | 11 | 11 | 3
  CO2, Month 5 | 0.3 (2.00) | -1.1 (2.07) | -1.0 (5.29)
  CO2, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  CO2, Follow-up | -0.3 (2.67) | -0.6 (1.86) | -0.6 (3.91)
  Glucose, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Glucose, Month 2 | -0.26 (1.087) | 0.46 (1.947) | 0.95 (1.622)
  Glucose, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Glucose, Month 5 | -0.85 (1.167) | -0.03 (1.698) | 1.70 (3.329)
  Glucose, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Glucose, Follow-up | -0.16 (1.315) | 0.22 (2.561) | 0.34 (1.354)
  Potassium, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Potassium, Month 2 | -0.01 (0.341) | -0.02 (0.251) | -0.20 (0.385)
  Potassium, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Potassium, Month 5 | 0.02 (0.544) | -0.11 (0.406) | -0.53 (0.404)
  Potassium, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Potassium, Follow-up | -0.06 (0.410) | -0.06 (0.277) | -0.44 (0.114)
  Sodium, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Sodium, Month 2 | 0.0 (1.81) | -1.0 (1.87) | 0.3 (2.25)
  Sodium, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Sodium, Month 5 | -0.6 (2.58) | -1.1 (0.94) | -2.7 (1.53)
  Sodium, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Sodium, Follow-up | -1.1 (2.77) | -1.2 (2.23) | -0.6 (0.55)
  Urea/BUN, Month 2: number analyzed (Participants) | 18 | 13 | 8
  Urea/BUN, Month 2 | -0.09 (1.417) | 0.12 (1.267) | 0.06 (1.130)
  Urea/BUN, Month 5: number analyzed (Participants) | 11 | 11 | 3
  Urea/BUN, Month 5 | 0.11 (0.905) | 0.67 (1.034) | -0.17 (0.764)
  Urea/BUN, Follow-up: number analyzed (Participants) | 16 | 11 | 5
  Urea/BUN, Follow-up | -0.36 (1.509) | 0.40 (1.059) | 1.00 (0.500)

9. Primary Outcome: Change From Baseline (Day 1) in Mean Corpuscular Volume (MCV) Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. MCV was recorded from Baseline up to Follow-up.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only those participants available at the time of assessment were analyzed
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Femtoliters
  Month 2: number analyzed (Participants) | 18 | 13 | 8
  Month 2 | 0.1 (2.07) | -0.2 (1.20) | -1.1 (1.24)
  Month 5: number analyzed (Participants) | 11 | 12 | 2
  Month 5 | 0.0 (1.95) | -0.6 (2.16) | -3.0 (0.00)
  Follow-up: number analyzed (Participants) | 16 | 12 | 4
  Follow-up | 0.2 (2.10) | 0.7 (1.20) | -2.8 (0.96)

10. Primary Outcome: Change From Baseline (Day 1) in Intra-ocular Pressure Assessment Over Period
Description: Change from Baseline is the value at indicated time point minus the Baseline value. Baseline measurement was recorded at Day 1. Intra-ocular pressure was recorded from Baseline up to Follow-up.
Time Frame: Baseline (Day 1) and approximately up to 6 months
Population: Safety population. Only those participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Millimeters of mercury
  Month 1: number analyzed (Participants) | 17 | 14 | 7
  Month 1 | 0.2 (3.47) | 0.7 (2.23) | 1.3 (2.98)
  Month 2: number analyzed (Participants) | 18 | 13 | 8
  Month 2 | 0.1 (3.46) | 1.2 (2.83) | 1.1 (3.18)
  Month 3: number analyzed (Participants) | 15 | 12 | 4
  Month 3 | -1.1 (4.07) | 0.7 (2.64) | 2.0 (4.69)
  Month 4: number analyzed (Participants) | 12 | 11 | 5
  Month 4 | -0.5 (2.35) | 1.2 (2.71) | 1.4 (5.86)
  Month 5: number analyzed (Participants) | 12 | 12 | 3
  Month 5 | -1.1 (3.60) | 1.2 (2.59) | -0.3 (5.77)
  Month Follow-up: number analyzed (Participants) | 16 | 13 | 6
  Month Follow-up | -1.3 (3.13) | 0.1 (2.72) | 0.7 (3.50)

11. Primary Outcome: Number of Participants With Blood Occult, Urine Glucose, Urine Ketones, and Urine Proteins by Dip Stick Analysis
Description: In this dipstick test, the level of blood occult and glucose, ketones, protein in urine samples were recorded as negative, trace, 1+, 2+, and 3+ (the plus sign increases with a higher level of glucose, ketones, or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive).
Time Frame: Approximately up to 6 months (up to follow-up)
Population: Safety population. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants
  Urine blood occult, Month 2, 1+: number analyzed (Participants) | 18 | 13 | 8
  Urine blood occult, Month 2, 1+ | 0 | 0 | 1
  Urine blood occult, Month 2, traces: number analyzed (Participants) | 18 | 13 | 8
  Urine blood occult, Month 2, traces | 3 | 2 | 0
  Urine blood occult, Month 5, traces: number analyzed (Participants) | 11 | 12 | 3
  Urine blood occult, Month 5, traces | 0 | 2 | 0
  Urine blood occult, Follow-up, traces: number analyzed (Participants) | 16 | 12 | 5
  Urine blood occult, Follow-up, traces | 1 | 0 | 0
  Urine glucose, Month 5, traces: number analyzed (Participants) | 11 | 12 | 3
  Urine glucose, Month 5, traces | 0 | 1 | 0
  Urine glucose, Follow-up, 1+ OR 1/4/G/DL (5%): number analyzed (Participants) | 16 | 12 | 5
  Urine glucose, Follow-up, 1+ OR 1/4/G/DL (5%) | 0 | 1 | 0
  Urine ketones, Month 2, traces: number analyzed (Participants) | 18 | 13 | 8
  Urine ketones, Month 2, traces | 1 | 0 | 0
  Urine ketones, Follow-up, traces: number analyzed (Participants) | 16 | 12 | 5
  Urine ketones, Follow-up, traces | 1 | 1 | 0
  Urine protein, Month 2, 1+: number analyzed (Participants) | 18 | 13 | 8
  Urine protein, Month 2, 1+ | 0 | 0 | 1
  Urine protein, Month 2, traces: number analyzed (Participants) | 18 | 13 | 8
  Urine protein, Month 2, traces | 3 | 0 | 0
  Urine protein, Month 5, 1+: number analyzed (Participants) | 11 | 12 | 3
  Urine protein, Month 5, 1+ | 0 | 1 | 1
  Urine protein, Follow-up, 1+: number analyzed (Participants) | 16 | 12 | 5
  Urine protein, Follow-up, 1+ | 0 | 1 | 0
  Urine protein, Follow-up, traces: number analyzed (Participants) | 16 | 12 | 5
  Urine protein, Follow-up, traces | 3 | 2 | 1

12. Primary Outcome: Number of Participants With Adverse Events (AEs)and Serious Adverse Events (SAEs)
Description: Number of participants with ocular and non-ocular AEs and SAEs were separately recorded. An AE is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. An SAE is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Time Frame: Approximately up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants
  Any AE, non-ocular | 11 | 9 | 3
  Any SAE, non-ocular | 2 | 0 | 0
  Any AE, ocular | 8 | 3 | 2
  Any SAE, ocular | 0 | 1 | 0

13. Primary Outcome: Number of Participants With Abnormal Visual Acuity of Potential Clinical Concern (PCI)
Description: Visual acuity was measured over 5 months and also during follow-up period. Visual acuity was measured using standardized early treatment of diabetic retinopathy study (ETDRS) visual acuity charts. Visual acuity measurement was performed by an examiner that had been appropriately trained. Screening, Month 2 and Month 5 data were considered as Best Corrected Visual Acuity (BCVA) data. A loss of greater than or equal to 15 letters in BCVA from Baseline was considered of PCI. Data for number of participants who met the criteria for PCI have been presented.
Time Frame: Approximately up to 6 months
Population: Safety population. Only those participants available at the time of assessment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 2 | 2 | 0

14. Primary Outcome: Number of Participants With Abnormal Pupil Examination of PCI
Description: Pupil abnormalities were of different types. Meibomian gland dysfunction was measured as obvious inspissation (debris). Mild injection, no trichiasis (lid thickening), or two step worsening was analyzed. Afferent pupillary defect, motility examination, PERRL, confrontation visual field was measured as a new definite abnormality. Left and right both eyes were examined.
Time Frame: Up to follow-up (approximately 6 months)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 2 | 1 | 1

15. Primary Outcome: Number of Participants With Abnormal Conjunctival Examination of PCI
Description: A two step worsening in the conjunctival examination was considered a value of PCI. Participants were analyzed for conjunctival examination up to follow-up (6 months).
Time Frame: Up to follow-up (approximately 6 months)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Abnormal Anterior Chamber Examination of PCI
Description: A two step worsening in the anterior chamber examination was considered a value of PCI. The participants were examined for any anterior chamber abnormality. Fibrinous response and obvious aqueous haze were considered abnormalities related to anterior chamber examination.
Time Frame: Approximately up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormal Corneal Examination of PCI
Description: A two step change in any of the lens opacity categories was categorized as of PCI. Corneal epithelium was defined as abnormal when punctate keratopathy was measured as mild, moderate, severe; epithelial edema was measured as subtle epithelial haze, mild patchy microcystic changes, diffuse microcystic changes, and/or investigator determined abnormality. Stromal opacity/ edema was measured by investigator when stroma identifies opacity or edema. Corneal staining was measured as obvious (<=20) localized or diffuse punctate staining areas, severe localized or diffuse punctate staining. Participants were analyzed for any of the mentioned abnormality over 6 weeks (up to follow-up period).
Time Frame: Approximately up to 6 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 2 | 0 | 0

18. Primary Outcome: Number of Participants With Abnormal Lens Opacity of PCI Using Age Related Eye Disease Study (AREDS) Scale
Description: A two step change in any of the lens opacity categories was considered a value of PCI. Aphakia (surgical removal of lens) or pseudophakia was noted if any. Stroma opacity or edema was measured by investigator when it was detected as edema or opacity in stroma.
Time Frame: Approximately up to 6 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 0 | 1 | 1

19. Primary Outcome: Number of Participants With Abnormal Tear Films of PCI
Description: Tear film abnormalities were based on the clinical judgment of investigator. Tear film thickness was analyzed and it was reported whether the film was increased or decreased or was normal. Presence of debris or mucus was also reported. Other test were tear lake analysis and checking of discharge from eyes.
Time Frame: Approximately up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 3 | 1 | 1

20. Primary Outcome: Number of Participants With Any Grade 2 Plus Worsening of Meibomian Gland Function
Description: Meibomian gland dysfunction was measured as obvious insipisation/debris, mild injection, no trichiasis or lid thickening; inspisation, debris, obvious injection, lid thickening, may have trsichiasis; or a two step worsening. Any 2+ worsening of Meibomian gland function was considered a value of PCI.
Time Frame: Approximately up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 1 | 0 | 1

21. Primary Outcome: Number of Participants With Abnormal (Dilated) Fundus Examination
Description: Dilation of fundus was examined post dosing up to 6 months. Number of participants with abnormal change from Baseline indicating dilation of fundus of eye was reported. Change from Baseline was the value at indicated time point minus the Baseline value. The abnormalities were posterior vitreous separation, pale optic nerve, fluid in the posterior pole, drusen, thick arterio-venous changes, pigment changes, cystoids, macular edema, drying of posterior fluid or sub-retinal fluid, underlying central atrophy, and retinal pigment epithelial changes etc. Refraction measurement were determined at the screening and 2 month/5 month visits in order to determine BCVA.
Time Frame: Approximately up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants | 4 | 1 | 2

22. Secondary Outcome: Change From Baseline (Screening Visit) in BCVA at Month 2 and 5
Description: Change from Baseline in BCVA is the value at indicated time point minus the Baseline value. BCVA at screening visit was used as statistical Baseline. Only data before post-dose intravitreal injection of Avastin/ Lucentis (IVT) has been presented. Arithmetic mean was presented as data values; however statistical analysis is based on means of observed case (OC) data. The screening was used as a Baseline visit that was within or at 14 days of Day 1. Screening visit BCVA values were used to perform statistical comparison at month 2 and 5.
Time Frame: From Baseline (screening visit), Month 2, and Month 5
Population: Efficacy population included all participants in safety population who have classic choroidal neovascularization present as detected by fluorescein angiography in the previous screening visit.
Measure: Mean (Standard Deviation); unit: Number of letters
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 13 | 12 | 4
Number of letters
  IVT Treatment naive, Month 2: number analyzed (Participants) | 8 | 7 | 3
  IVT Treatment naive, Month 2 | 0.1 (4.85) | -5.3 (6.24) | -0.7 (3.06)
  IVT Treatment naive, Month 5: number analyzed (Participants) | 5 | 7 | 1
  IVT Treatment naive, Month 5 | -5.6 (12.60) | -5.3 (6.70) | -3.0 (NA) — Since only 1 participant was analyzed, SD will not be applicable.
  Previously treated with IVT, Month 2: number analyzed (Participants) | 5 | 4 | 0
  Previously treated with IVT, Month 2 | -1.6 (4.28) | -3.5 (4.65) |
  Previously treated with IVT, Month 5: number analyzed (Participants) | 4 | 3 | 0
  Previously treated with IVT, Month 5 | -1.3 (3.30) | -2.0 (7.21) |
Statistical Analysis 1: Comparison: 5 mg/mL TID; Month 2 versus screening visit; Test type: Superiority; ANCOVA — Analysis of covariance (ANCOVA) model was used to perform statistical analysis based on treatment, visit, fixed effect terms etc; Mean Difference (Net) = -0.43, 95% CI 2-sided [-3.18 to 2.31], Standard Error of Mean 1.362
Statistical Analysis 2: Comparison: 5 mg/mL TID; Month 5 versus screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 22, analysis 1]; Mean Difference (Net) = -3.80, 95% CI 2-sided [-7.13 to -0.46], Standard Error of Mean 1.659
Statistical Analysis 3: Comparison: 2 mg/mL TID; Month 2 versus screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 22, analysis 1]; Mean Difference (Net) = -4.15, 95% CI 2-sided [-7.52 to -0.78], Standard Error of Mean 1.672
Statistical Analysis 4: Comparison: 2 mg/mL TID; Month 5 versus screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 22, analysis 1]; Mean Difference (Net) = -4.03, 95% CI 2-sided [-7.53 to 0.53], Standard Error of Mean 1.740

23. Secondary Outcome: Change From Baseline (Screening Visit) in Optical Coherence Tomography (OCT) Central Subfield Over 5 Months
Description: The OCT effect is a pharmacodynamics (PD) measure of daily repeated dosing of Pazopanib. The anatomic effects of pazopanib treatment were limited to investigator determined assessment of OCT central subfield retinal thickness due to heterogeneity of participant population and the low likelihood of utility of central reading center determination. The OCT equipment used was approved by central OTC reading center. OCT scans were collected at indicated time points and were evaluated by Investigator. Thus, grading of further secondary objectives was not performed as per the study team. Change from Baseline is the value at indicated time point minus the Baseline value. The screening was used as a Baseline visit that was within or at 14 days of Day 1. Screening visit BCVA values were used to perform statistical comparison at month 2 and 5.
Time Frame: From Baseline (Screening visit) and up to 5 months
Population: Pharmacodynamic subpopulation included participants that were analyzed for PD outcome measures. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 13 | 12 | 4
Microns
  Treatment naive, Month 1: number analyzed (Participants) | 8 | 7 | 3
  Treatment naive, Month 1 | 8.3 (48.19) | 41.1 (99.51) | -18.0 (37.40)
  Treatment naive, Month 2: number analyzed (Participants) | 8 | 7 | 3
  Treatment naive, Month 2 | 16.3 (62.32) | 18.3 (45.09) | 3.0 (47.32)
  Treatment naive, Month 3: number analyzed (Participants) | 6 | 7 | 2
  Treatment naive, Month 3 | -31.3 (43.43) | 31.3 (61.36) | 12.0 (5.66)
  Treatment naive, Month 4: number analyzed (Participants) | 5 | 6 | 2
  Treatment naive, Month 4 | -19.2 (52.77) | -15.3 (41.28) | -168.5 (246.78)
  Treatment naive, Month 5: number analyzed (Participants) | 5 | 7 | 1
  Treatment naive, Month 5 | -15.6 (52.13) | 7.3 (45.11) | 16.0 (NA) — No SD can be calculated for one participant analyzed.
  Previously treated, Month 1: number analyzed (Participants) | 5 | 4 | 1
  Previously treated, Month 1 | 46.4 (130.30) | -1.3 (27.93) | 36.0 (NA) — No SD can be calculated for one participant analyzed.
  Previously treated, Month 2: number analyzed (Participants) | 5 | 4 | 0
  Previously treated, Month 2 | -99.0 (180.74) | -10.0 (108.19) |
  Previously treated, Month 3: number analyzed (Participants) | 5 | 3 | 0
  Previously treated, Month 3 | -66.2 (126.35) | 2.0 (37.99) |
  Previously treated, Month 4: number analyzed (Participants) | 4 | 3 | 0
  Previously treated, Month 4 | -86.8 (151.02) | 0.3 (87.37) |
  Previously treated, Month 5: number analyzed (Participants) | 4 | 3 | 0
  Previously treated, Month 5 | -55.5 (159.53) | 3.0 (66.43) |
Statistical Analysis 1: Comparison: 5 mg/mL TID; For Month 1 versus Screening visit; Test type: Superiority; ANCOVA — ANCOVA model was used to perform statistical analysis based on treatment, visit, fixed effect terms, Baseline OCT central subfield as covariate, and participant within treatment as a random effect term; Mean Difference (Net) = 8.28, 95% CI 2-sided [-25.72 to 42.29], Standard Error of Mean 16.899
Statistical Analysis 2: Comparison: 5 mg/mL TID; Month 2 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -1.21, 95% CI 2-sided [-35.73 to 33.31], Standard Error of Mean 17.177
Statistical Analysis 3: Comparison: 5 mg/mL TID; Month 3 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -5.11, 95% CI 2-sided [-41.08 to 30.86], Standard Error of Mean 17.958
Statistical Analysis 4: Comparison: 5 mg/mL TID; Month 4 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -9.92, 95% CI 2-sided [-47.83 to 28.00], Standard Error of Mean 18.996
Statistical Analysis 5: Comparison: 5 mg/mL TID; Month 5 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = 2.42, 95% CI 2-sided [-35.50 to 40.33], Standard Error of Mean 18.996
Statistical Analysis 6: Comparison: 2 mg/mL TID; Month 1 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = 9.05, 95% CI 2-sided [-33.09 to 51.20], Standard Error of Mean 20.931
Statistical Analysis 7: Comparison: 2 mg/mL TID; Month 2 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -1.24, 95% CI 2-sided [-44.05 to 41.57], Standard Error of Mean 21.290
Statistical Analysis 8: Comparison: 2 mg/mL TID; Month 3 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = 15.39, 95% CI 2-sided [-28.28 to 59.06], Standard Error of Mean 21.757
Statistical Analysis 9: Comparison: 2 mg/mL TID; Month 4 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -16.82, 95% CI 2-sided [-61.28 to 27.63], Standard Error of Mean 22.183
Statistical Analysis 10: Comparison: 2 mg/mL TID; Month 5 versus Screening visit; Test type: Superiority; ANCOVA — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Net) = -2.16, 95% CI 2-sided [-45.83 to 41.51], Standard Error of Mean 21.757

24. Secondary Outcome: Change in Neo-vascular Size and Lesion Size Over Period
Description: The analysis was planned to be performed up to 6 months; however, due to heterogeneity of the population and the low likelihood of the utility of the data, the anatomic effects of the pazopanib treatment in this treatment were limited to investigator determined assessment of OCT central subfield retinal thickness. Thus, the study team decided not to have DARC (central reading center) perform the grading for the secondary PD outcomes like lesion size and change with respect to time were not analyzed. Thus, data was not collected for this outcome measure.
Time Frame: Up to 6 weeks
Population: PD population was planned for analysis of this outcome; however, Data was not collected for this outcome measure.
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Lesion Types Over Period
Description: Number of participants with type of lesion were reported as determined by Investigator. Occult and minimally classic were the two types of lesions reported.
Time Frame: Up to 6 months
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
Number analyzed (Participants) | 19 | 15 | 8
Participants
  Occult | 16 | 11 | 3
  Minimally classic | 2 | 4 | 5

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected approximately up to 6 months
Description: Safety Population was used to collect AE and SAE data
Arm/Group | 5 mg/mL TID | 2 mg/mL TID | 5 mg/mL QD
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/15 | 0/8
Other Adverse Events (participants affected / at risk) | 15/19 | 9/15 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg/mL TID (N=19) | 2 mg/mL TID (N=15) | 5 mg/mL QD (N=8)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5 mg/mL TID (N=19) | 2 mg/mL TID (N=15) | 5 mg/mL QD (N=8)
Eye pain (Eye disorders) | 2 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 1 | 0
Macular degeneration (Eye disorders) | 1 | 1 | 0
Retinal disorder (Eye disorders) | 2 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Optic disc haemorrhage (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Posterior capsule opacification (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Sensation of foreign body (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.